CLINICAL TRIAL: NCT05065320
Title: Tools for the Integrated Management of Childhood Illness: Evaluation of Pulse Oximetry and Clinical Decision Support Algorithms in Primary Care. Cross-country Quasi-experimental Pre-post Study, With Embedded Mixed Methods Studies, Cost and Modelled Cost-effectiveness in Kenya and Senegal
Brief Title: Tools for the Integrated Management of Childhood Illness: Cross-country Quasi-experimental Pre-post Study in Kenya and Senegal
Acronym: TIMCI
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: PATH (Other); University of Nairobi (Other); Cheikh Anta Diop University, Senegal (Other); Burnet Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ERC.0003406
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-11

CONDITIONS: Childhood Severe Illness; Pneumonia; Primary Health Care; Hypoxia; Referreal and Consultation; Decision Support Systems, Clinical; Oxymetry
MeSH Terms: conditions — Pneumonia; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By introducing pulse oximetry, with or without clinical decision support algorithms, to primary care facilities in India, Kenya, Senegal and Tanzania, the Tools for Integrated Management of Childhood Illness (TIMCI) project aims to contribute to reducing morbidity and mortality for sick children under-five while supporting the rational and efficient use of diagnostics and medicines by healthcare providers.

The multi-country, multi-method evaluation aims to generate evidence on the health and quality of care impact, operational priorities, cost and cost-effectiveness of introducing these tools to facilitate national and international decision-making on scale-up.

DETAILED DESCRIPTION:
This registry entry describes the quasi-experimental pre-post studies conducted in Kenya and Senegal. In India and Tanzania, pragmatic cluster randomised controlled trials (RCTs) are conducted (NCT04910750). These studies evaluating health, clinical and quality of care impact are complemented by embedded multi-method studies in all countries, including modified Service Provision Assessments, facility-based process mapping and time-flow studies, in-depth interviews (IDIs) with caregivers and healthcare providers, online key stakeholder surveys and key informant interviews, routine data review, and an economic evaluation.

We enrol sick children 0 to 59 months of age attending government primary care facilities in before and after implementation of pulse oximetry and CDSA. Interventions are implemented with a package of training on the use of devices and refresher IMCI, supportive supervision, operational support and community engagement.

As part of the intervention, facilities are provided with handheld, UNICEF-approved, pulse oximeters along with guidance and training for healthcare providers. In Senegal, healthcare providers are advised to measure oxygen saturation (SpO2) on all children under 2 months of age, all children 2 to 59 months of age with cough or difficulty breathing or with signs of moderate or severe disease based on Integrated Management of Childhood Illness (IMCI); in Kenya, healthcare providers are advised to measure oxygen saturation for all sick children. Providers are advised to urgently refer children with SpO2 <90% in Kenya and <92% in Senegal. The tablet-based CDSA provides step-by-step support to healthcare providers through consultations, providing national guideline-based recommendations on assessment, diagnosis and treatment based tailored to the individual child based on information entered by the provider. Following training, providers are advised to use CDSA for all consultations with sick children under 5 years of age.

Sociodemographic and clinical data are collected from caregivers and records of enrolled sick children at study facilities, with phone follow-up on Day 7. Two primary outcomes are assessed for the quasi-experimental pre-post study: referrals to a higher level of care at Day 0 consultation; and antibiotic prescriptions on Day 0. These reflect the aim that the intervention increases detection of severe disease, and therefore increasing referral, whilst promoting antimicrobial stewardship, and therefore reducing antibiotic prescription. Secondary outcomes, relating to hypoxaemia, hospitalisation, referral, antimicrobial prescription, follow-up, health status are further detailed in the attached full protocol and statistical analysis plan available.

The pre-post study sample size was originally estimated for a planned 15 month study, with 3 months pre- (Q1) and 12 months post-intervention (Q2-5), with comparison of Q1 and Q5 for the primary outcome. Calculations were based on detecting a ≥50% increase in Day 0 referrals (from 3%, based on DHIS2, SPA and facility estimates), with 80% power, 0.05 alpha and ICC of 0.00547. A relatively large detectable difference was chosen given that a relatively high proportion of referrals may not be completed.5 46 Day 0 referrals, rather than antibiotic prescriptions (with baseline estimated at 60% with ICC 0.05), drove the sample size calculation. We estimated needing 17 facilities, recruiting an average of 690 children per facility per 3-month period in Kenya, and 18 facilities recruiting 510 children per facility per period in Senegal.

Following lower than anticipated recruitment in the baseline of the pre-post study, sample size was re-evaluated resulting in a decision to add two facilities per country, extend the baseline (to 6-7 months), and reduce the post-intervention period (to 9-10 months). A minimum of 7429 and 6760 children were estimated to be needed in each period in Kenya and Senegal respectively, with recruitment continuing after meeting the minimum sample size in order to allow for description of changes over time and with overlapping seasonal periods, in line with the intention of the original design.

Study approval has been granted by all relevant institutional review boards, national and WHO ethical review committees. Findings will be shared with communities, healthcare providers, Ministries of Health and other local, national and international stakeholders to facilitate evidence-based decision-making on scale-up.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-59 months of age for whom caregivers provide consent
* Consulting for an illness, or reported to be unwell when attending for a routine visit (e.g. vaccination, growth or chronic disease monitoring)

Exclusion Criteria:

* Children in the immediate post-natal period or first day of life
* Attending for a consultation related to trauma only (including new and follow-up presentations for burns, injuries, wounds)
* Admitted within an inpatient part of the facility (including neonates delivered at the facility admitted with their mother)
* Enrolled in the study within the preceding 28 days at any study facility

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 0 - 59 months, for whom caregivers provide consent, will be eligible if attending any study facility with an illness, excluding those admitted as inpatients within the facility, or attending for a consultation related to trauma only.
Sampling Method: Probability Sample
Enrollment: 51590 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of children referred by a primary care healthcare provider to a higher level of care (either to a hospital or to an inpatient part of a larger primary healthcare facility) at Day 0 consultation | At time of enrolment
  The denominator will be all children recruited. Only urgent referrals will be considered.
Proportion of children prescribed an antibiotic at Day 0 | At time of enrolment
  Only antibacterials for systemic use will be taken into account for the definition of antibiotics. All children recruited will be counted in the denominator.

SECONDARY OUTCOMES:
Proportion of children with a severe complication (death or secondary hospitalisation) by Day 7 | From enrolment up to 7 days after
  Secondary hospitalisation refers to any delayed hospitalisation (occurring at any point greater than 24 hours after Day 0 consultation) and any hospitalisation occurring without referral. The denominator is all enrolled children..
Proportion of children admitted to hospital within 24 hours of the Day 0 primary care consultation and as a result of a referral | From enrolment up to 1 day after
  This is used as a proxy for 'appropriate referral' of children, as those with severe disease should generally be admitted to hospital. The denominator for this outcome is also all children enrolled in the study, rather than only referred children. This is because the proportion of referred children that are admitted may be high in routine care, in the context of an inappropriately low referral rate. The aim of the intervention is therefore to increase the overall referral rate of children with severe disease. Hospital admission is chosen as the proxy of severe disease rather than using primary care classification of severe disease, as there are inadequacies in the classification of severe disease in routine practice. A child will be considered admitted to hospital 24hrs of Day0 consultation if the date of hospitalization is the same as Day0 date or is one day after Day0 date.
Proportion of children who completed referral, as reported at day 7 follow-up | From enrolment up to 10 days after
  Only urgent referrals will be considered. A referral will be considered completed if a child attended a hospital, whether was admitted or not. A window of +3 days from Day 7 is considered.
Proportion of children cured (defined as caregiver reported recovery from illness) by Day 7 | From enrolment up to 10 days after
  The denominator will be all children recruited. A window of +3 days from Day 7 is considered.
Proportion of children with non-severe disease referred to a higher level of care on Day 0 | At time of enrolment
  Only urgent referrals will be considered. Only urgent referrals will be considered.
Average length of stay (in days) of children admitted to hospital | From hospital admission to discharge
  If a child is hospitalised twice, the first hospitalization will be used and second hospitalizations will be reported separately. The denominator will be all hospitalised children. This is not a time-to-event outcome measure, as it will be analysed as a continuous variable.
Proportion of children prescribed a diagnosis-appropriate antibiotic | At time of enrolment
  Appropriateness of antibiotic prescription in relation to diagnosis will be evaluated as:
  * diagnosis for which a systemic antibiotic was indicated and a systemic antibiotic was prescribed
  * diagnosis for which a systemic antibiotic was not indicated and systemic antibiotic was prescribed
  * first-line (or second-line) antibiotics were prescribed according to recommendations for IMCI diagnoses for which specific antibiotic(s)are indicated Diagnoses will be classified according to whether systemic antibiotics are indicated, based on IMCI and other relevant national guidelines as used for the CDSA.
Proportion of febrile children tested for malaria at Day 0 | At time of enrolment
  A child will be considered to be febrile if history of fever was reported by the caregiver before the consultation or temperature was recorded to be above or equal 37.5 C°. Only febrile children will be counted in the denominator.
Proportion of malaria positive children prescribed an antimalarial | At time of enrolment
  Only children with a positive malaria test result will be counted in the denominator.
Proportion of malaria negative children prescribed an antimalarial | At time of enrolment
  Only children with a negative malaria test result will be counted in the denominator.
Proportion of untested children prescribed an antimalarial | At time of enrolment
  Only children untested for malaria will be counted in the denominator.
Proportion of children with severe, moderate and mild hypoxaemia, adjusted for sites at high altitude | At time of enrolment
  The following SpO2 values ranges will be used: SpO2 < 90%, 90% ≤ SpO2 < 92% and 92% ≤ SpO2 < 94%. All children recruited will be in the denominator.
Proportion of children with hypoxaemia (according to differing cut-offs) with severe complication | At time of enrolment
  The following SpO2 values ranges will be used: SpO2 < 90%, 90% ≤ SpO2 < 92% and 92% ≤ SpO2 < 94%, spurious values and missing values. Each SpO2 group will be the denominator of each proportion.
Proportion of children with severe hypoxaemia not meeting any other clinical criteria for severe disease | At time of enrolment
  Country's specific cut-off for severe hypoxaemia will be used. All children recruited will be in the denominator.
Proportion of children referred with hypoxaemia who receive oxygen at hospital | At time of enrolment and at time of hospitalization
  All children recruited will be in the denominator. Referral and hypoxaemia are assessed at Day0 consultation. Oxygen use at hospital is only available for hospitalised children from hospital records. At the time of enrolment hypoxaemia is measured and referral advise might be issued. Whether the child received oxygen or not at hospital is evaluated based on hospital registry and it refers to oxygen given at arrival to hospital. The specified time frame takes into account that the outcome is evaluated considering information recorded at different time points.
Proportion of children attending scheduled follow-up at the same facility by Day 7 | From enrolment up to 7 days after
  All children recruited will be in the denominator.
Proportion of children presenting for unscheduled follow-up to any health facility by Day 7 | From enrolment up to 7 days after
  All children recruited will be in the denominator.

CONTACTS AND LOCATIONS:
Overall Officials: Kaspar Wyss, Prof, PhD, Principal Investigator — Swiss Tropical & Public Health Institute; Valérie D'Acremont, MD, PhD, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (2):
- University of Nairobi, Nairobi, Kenya
- UCAD, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared that underlie the quasi-experimental pre-post study outcomes as described in the study protocol, after anonymisation.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data will be available immediately following the cross-country publication of the quasi-experimental pre-post study outcomes. No end date.
Access Criteria: Anyone who wishes to access the data. Data will be available indefinitely on the TIMCI project space on Zenodo.
URL: https://zenodo.org/communities/timci

REFERENCES:
- [Derived] Langet H, Faye PM, Njiri F, Cicconi S, Levine GA, Glass TR, Kosgei RJ, Ngari K, Schaer F, Thiongane A, Tine JAD, Ba M, Bohle LF, Emmanuel-Fabula M, Faye MM, Horton S, Miheso A, Mugo M, Ngutu M, Ruffo M, Shauri J, Sougou NM, D'Acremont V, Wyss K, Ndiaye O, Beynon F; TIMCI Collaborator Group. Effectiveness of introducing pulse oximetry and clinical decision support algorithms for the management of sick children in primary care in Kenya and Senegal on referral and antibiotic prescription: the TIMCI quasi-experimental pre-post study. EClinicalMedicine. 2025 May 12;83:103196. doi: 10.1016/j.eclinm.2025.103196. eCollection 2025 May. PMID 40474998
- [Derived] Beynon F, Langet H, Bohle LF, Awasthi S, Ndiaye O, Machoki M'Imunya J, Masanja H, Horton S, Ba M, Cicconi S, Emmanuel-Fabula M, Faye PM, Glass TR, Keitel K, Kumar D, Kumar G, Levine GA, Matata L, Mhalu G, Miheso A, Mjungu D, Njiri F, Reus E, Ruffo M, Schar F, Sharma K, Storey HL, Masanja I, Wyss K, D'Acremont V; TIMCI Collaborator Group. The Tools for Integrated Management of Childhood Illness (TIMCI) study protocol: a multi-country mixed-method evaluation of pulse oximetry and clinical decision support algorithms. Glob Health Action. 2024 Dec 31;17(1):2326253. doi: 10.1080/16549716.2024.2326253. Epub 2024 Apr 29. PMID 38683158

DOCUMENTS (3):
  • Study Protocol (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT05065320/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT05065320/SAP_001.pdf
  • Informed Consent Form (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT05065320/ICF_002.pdf